CLINICAL TRIAL: NCT06246955
Title: "Live Fully With Cancer": Assessing the Impact of an Acceptance and Commitment Therapy and Compassion-Based Virtual Group Intervention for Diverse Cancer Patients
Brief Title: Acceptance and Commitment Therapy and Compassion-Based Virtual Group Therapy to Improve Psychological Wellbeing in Patients With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-005161; NCI-2024-00399 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-005161 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (group therapy sessions) (Experimental): Patients attend acceptance and commitment virtual group therapy sessions over 1.5 hours each, once a week for 6 weeks.
  Interventions: Behavioral: Behavioral Intervention: Group Therapy Session; Other: Survey Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention: Group Therapy Session — Attend virtual group therapy sessions
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
Other: Survey Administration — Ancillary study

SUMMARY:
This clinical trial tests how well acceptance and commitment therapy and compassion based virtual group therapy works to improve psychological wellbeing, such as compassion, understanding, and flexibility, in patients with cancer. Receiving a cancer diagnosis, undergoing cancer treatment, and living with cancer- or treatment-related symptoms have often been found to be associated with elevated distress and decreased quality of life for individuals, even when the disease is stable or in remission. Acceptance and Commitment Therapy (ACT) has demonstrated considerable benefits on individuals' quality of life, psychological flexibility, and amelioration of psychological distress following a cancer diagnosis and in the face of uncertainty, loss, and challenges associated with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess if participants perceive compassion and understanding by the provider who facilitates the virtual group intervention.

II. To assess if participation in the ACT-based group intervention is associated with increases in patients' self-reported psychological flexibility as well as amelioration in psychological and physical distress.

SECONDARY OBJECTIVE:

I. To assess if participation in the ACT-based group intervention is associated with increases in patients' self-reported mindfulness, self-compassion, meaning and purpose, and posttraumatic growth.

OUTLINE:

Patients attend acceptance and commitment virtual group therapy sessions over 1.5 hours each, once a week for 6 weeks.

After completion of study treatment, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Being an adult (18 years or older)
* Being a patient of Mayo Clinic Arizona
* Having a cancer diagnosis, having treatment planning in progress, undergoing cancer-related treatment, or having completed cancer within the past 2 years (in recent survivorship
* Experiencing stress or challenges related to cancer and having treatment goals that align with the purpose of the group
* Having self reported proficiency to read/write/speak English
* Expressing interest and commitment to attend all six virtual group sessions

Exclusion Criteria:

* Patients' inability to take part in and benefit from the virtual group therapy based on clinical judgment of the psychosocial oncology team member who completes the psychosocial evaluation, which may include having active suicidal or homicidal intent, experiencing uncontrolled psychotic symptoms, having untreated personality disorder/characteristics that are likely disturbing in a group setting, and/or having moderate to severe cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Participant perceived compassion and understanding by the group therapy provider - SCQ | From baseline to 1 month post session 6
  Will be assessed based on average scores using the 5-item Sinclair Compassion Questionnaire (SCQ), answered using a 5-point scale (strongly disagree, disagree, neutral, agree, strongly agree)
Patients' self-reported psychological flexibility - COMPACT-15 | From baseline to 1 month post session 6
  Will be assessed using the 15-item Comprehensive Assessment of Acceptance and Commitment Therapy Processes (COMPACT-15). Questions are answered on a scale of 0-6 (strongly disagree, moderately disagree, slightly disagree, neither agree nor disagree, slightly agree, moderately agree, strongly agree).
Patients' self-reported psychological flexibility - Psy-Flex | From baseline to 1 month post session 6
  Will be assessed using the 6-item Psy-Flex scale. Questions are answered on a 5-point scale (very often, often, from time to time, seldom, very seldom) based on experiences over the past 7 days.
Physician and psychological distress - PROMIS-29 | From baseline to 1 month post session 6
  Will be assessed using the Patient Reported Outcomes Measurement Information System (PROMIS)-29 v2.0 Profile, which assesses pain intensity using a 0-10 numeric rating scale across seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance), with four items per domain.

SECONDARY OUTCOMES:
Self reported mindfulness | Baseline; 1 month post session 6 (not assessed at mid-group to reduce patient survey burden)
  Will be assessed using the 15-item Five Facet Mindfulness Questionnaire - Short Form (FFMQ-SF). Questions are answered on a scale of 1-5 (1-never or very rarely true, 2-rarely true, 3-sometimes true, 4-often true, 5-very often or always true).
Self-compassion | Baseline; 1 month post session 6 (not assessed at mid-group to reduce patient survey burden)
  Will be assessed using the the 12- item Self-Compassion Scale Short Form (SCS-SF). Questions are answered on a scale of 1-5 where 1 = almost never and 5 = almost always.
Meaning and purpose | Baseline; 1 month post session 6 (not assessed at mid-group to reduce patient survey burden)
  Will be assessed using the 5-item Presence of Meaning subscale of the Meaning in Life Questionnaire (MLQ). Questions are answered on a 7-point scale (absolutely untrue, mostly untrue, somewhat untrue, cannot say true or false, somewhat true, mostly true, absolutely true).
Posttraumatic growth | Baseline; 1 month post session 6 (not assessed at mid-group to reduce patient survey burden)
  Will be assessed using the 10-item Posttraumatic Growth Inventory - Short Form (PTGI-SF). Questions are answered on a scale of 0-5 where 0 = I did not experience this change following my cancer diagnosis; 1 = I experienced this change to a very small degree following my cancer diagnosis; 2 = I experienced this change to a small degree following my cancer diagnosis; 3 = I experienced this change to a moderate degree following my cancer diagnosis; 4 = I experienced this change to a great degree following my cancer diagnosis; and 5 = I experienced this change to a very great degree following my cancer diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Tao, PhD, LP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials